CLINICAL TRIAL: NCT00091078
Title: A Phase IIA Study to Determine the Safety and Efficacy of A NCI-Supplied Agent: G3139 (NSC 683428, IND 58842) and Imatinib Mesylate in Patients With Refractory or Relapsed Gastrointestinal Stromal Tumor
Brief Title: Oblimersen and Imatinib Mesylate in Treating Patients With Advanced Gastrointestinal Stromal Tumors That Cannot Be Removed By Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02883; 2003-0761; 6122; N01CM62202 (NIH)
Record Dates: First submitted 2004-09-07; First posted 2004-09-08 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Gastrointestinal Stromal Tumor
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — oblimersen; Imatinib Mesylate

ARMS (1):
- Treatment (oblimersen sodium and imatinib mesylate) (Experimental): Patients receive oblimersen IV continuously on days 1-14. Patients also receive oral imatinib mesylate on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: oblimersen sodium; Drug: imatinib mesylate; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: oblimersen sodium — Given IV
  Other Names: augmerosen; G3139; G3139 bcl-2 antisense oligodeoxynucleotide; Genasense
Drug: imatinib mesylate — Given orally
  Other Names: CGP 57148; Gleevec; Glivec
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Imatinib mesylate may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Oblimersen may help imatinib mesylate kill more tumor cells by making tumor cells more sensitive to the drug. This phase II trial is studying how well giving imatinib mesylate together with oblimersen works in treating patients with advanced gastrointestinal stromal tumor that cannot be removed by surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy of G3139 (bcl-2 antisense oligonucleotide) plus imatinib mesylate in GIST patients with limited or generalized progression after therapy with imatinib.

II. To assess the safety of G3139 plus imatinib mesylate in GIST patients with limited or generalized progression after therapy with imatinib.

III. To determine whether expression of BCL-2 correlates with survival, time to progression or response rate in patients with GIST treated with G3139 plus imatinib.

OUTLINE: This is a multicenter study. Patients are stratified according to extent of disease progression (limited vs generalized).

Patients receive oblimersen IV continuously on days 1-14. Patients also receive oral imatinib mesylate on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed for survival.

PROJECTED ACCRUAL: A total of 96 patients (48 per stratum) will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* A pre-imatinib paraffin block of tumor or 20 unstained slides should be submitted for correlative studies if available
* All patients must have either "limited" progression on imatinib (arm 1, some but not all tumor foci progressing and are not amenable to local therapy) or "generalized" progression (arm 2, widespread progression of all tumor foci) after adequate therapy with imatinib mesylate (> or = 400 mg/day for at least 6 weeks)
* Histologically confirmed diagnosis of Kit-expressing advanced GIST; advanced GIST is defined by patients who have disease that is unresectable; this includes patients with metastatic disease or primary tumors that cannot be safely removed by a sarcoma surgical oncologist
* Measurable disease by CT; tests used to assess disease must be done within 28 days prior to registration. If a targeted lesion has been previously embolized or irradiated, or if the patient has received imatinib, there must be objective evidence of progression to be considered for response assessment
* ECOG performance status 0-2
* At least 4 weeks and recovery from effects of prior therapy (i.e radiation, biotherapy, chemotherapy other than imatinib mesylate, or embolization;) recovery from the effects of prior therapy such that they are less than or equal to grade 1 in severity for non-hematological toxicities excluding nausea and vomiting controlled with standard anti-emetic regimens, alopecia, fatigue, and peripheral edema
* Absolute neutrophil count (ANC) >= 1000/mm3
* Platelets >= 100,000/mm3
* Serum creatinine =< 1.5 x ULN
* Serum bilirubin =< 1.5 x ULN
* Serum SGOT or SGPT =< 2.5 x ULN if no liver metastases or =< 5 x ULN if liver metastases are present
* PT and PTT =< 1.5 x ULN
* Understand and sign written informed consent in accordance with institutional and federal guidelines
* All patients must have progressive disease defined as 1) an increase in unidimensional tumor size of > or = 10% AND did not meet criteria for PR by CT density, 2) any new lesions, including new tumor nodules in a previous cystic tumor
* Patients with widespread metastatic and progressive disease will be eligible for this protocol
* Patients without widespread metastases will be evaluated by a sarcoma surgical oncologist to determine the benefit of and risk of surgical resection; if surgical resection is not recommended, the patient will be eligible for therapy with the study drug
* Pregnancy or lactation; women or men of reproductive potential must agree to use an effective barrier contraceptive method during treatment and for three months after the last dose of drug; women of reproductive potential must have a negative serum pregnancy test within 7 days prior to registration; post-menopausal women must be amenorrheic for at least 12 months to be considered of non-child bearing potential

Exclusion Criteria:

* Significant concurrent medical disease other than cancer including:

  * New York Heart Association class III or IV cardiac problems (e.g., congestive heart failure, acute myocardial infarction within 2 months of study)
  * Uncontrolled chronic renal or liver disease
  * Uncontrolled diabetes
  * Uncontrolled seizure disorder
  * Active uncontrolled infection, e.g., HIV
  * Organ allografts
* History of second cancer, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for 5 or more years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2005-09; Primary Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Response defined using the Choi criteria | 2 months
  The design method of Thall, Simon and Estey will be used.
Toxicity defined as any of the following events: regimen-related death, transaminitis, infection, or leukopenia grade 3 or higher using NCI CTCAE version 3.0 | 2 months
  The design of Thall, Simon and Estey will be used.

SECONDARY OUTCOMES:
Disease-free survival | Up to 4 years
  Regression analyses will be performed to assess the ability of patient prognostic factors to predict these time-to-event outcomes (survival analyses), as well as the probabilities of response and toxicity (logistic or extended logistic regression analyses).
Overall survival | Up to 4 years
  Regression analyses will be performed to assess the ability of patient prognostic factors to predict these time-to-event outcomes (survival analyses), as well as the probabilities of response and toxicity (logistic or extended logistic regression analyses).

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Trent, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States